CLINICAL TRIAL: NCT03668132
Title: The Language Functional Reorganization Following Subcortical Cerebral Infarction: A Longitudinal fMRI Study
Brief Title: Language Functional Reorganization in Subcortical Infarction Patients
Status: Completed | Type: Observational
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Yan Liu, Director of cerebrovascular department, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: LY-89514138
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Subcortical Aphasia; Ischemic Stroke
Keywords: Aphasia; Functional magnetic resonance imaging; Subcortical aphasia; Post-stroke aphasia; Cortical activation
MeSH Terms: conditions — Ischemic Stroke; Aphasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Left damage: Have the ischemic brain damage and the location of the damage ,and in the left brain
  Interventions: Other: ischemic brain damage
- Right damage: Have the ischemic brain damage and the location of the damage ,and in the right brain
  Interventions: Other: ischemic brain damage
- Normal control: Not have the ischemic brain damage
  Interventions: Other: ischemic brain damage

INTERVENTIONS:
Other: ischemic brain damage — Have or not have the ischemic brain damage and the location of the damage

SUMMARY:
Post stroke aphasia (PSA) is one of the most frequently happened deficiency of stoke, affecting speaking,comprehension, writing and reading of language. Generally, PSA is commonly seen in cortical damage, but in recent years it has been found that subcortical injury is also an important cause of PSA, which is called subcortical aphasia. Using fMRI technology, the investigators aim to investigate the language function of patients with subcortical cerebral infarction at different stages of recovery , and explored the mechanism of post-injury language reorganization in the brain.

The investigators recruited 60 first-episode acute cerebral infarction patients with one-side lesion in subcortical white matter (40 with left injury and 20with right injury) and 20 health volunteers. All participants are right-handed, and screened with MMSE, HAMD and HAMA to exclude cases of psychosis, post-stroke dementia and depression. Each participant was arranged to have three test sessions at different stages after the infarction (T1:within 3 days after onset of the stroke ; T2:28 ±3days after onset; T3: 90±3days after onset), with fMRI and Western aphasia battery (WAB) in each session.

The purpose of this study is to explore the pathogenesis of subcortical aphasia, and to understand the dynamic reorganization of language network during the recovery of language function.

DETAILED DESCRIPTION:
The participants were recruited from inpatients with acute ischemic stroke in Department of Cerebrovascular disease, The Guangzhou General Hospital of Guangzhou Military Command. The diagnose of ischemic stroke was made using the diagnostic criteria of the International Association of Neurological Diseases and Stroke Association in 1982. The classification criterias for ischemic stroke were based on the current international TOAST etiological classification method.

The study passed the approval of the ethics committee of General Hospital of Guangzhou Military Command , and all participants or their guardian signed informed consent. According to the location and diagnostic criteria, the participants were divided into three groups: left hemisphere infarction patients group ,right hemisphere infarction patients group and normal healthy control group. The participants performed 3 language functional behavior tests and functional magnetic resonance (fMRI) tests within3 days,28 ±3days ,90±3days after the onset of cerebral infarction. In the healthy control group, the above examination was performed only 1 times. Language functional behavioral assessments included the Chinese version of Western Aphasia Battery(WAB), spontaneous language frequency test(SLFT) and picture naming test(PNT). Examines of fMRI included task-state fMRI , resting-state fMRI and diffusion tensor imaging(DTI).

Task state function magnetic resonance design：Using the block design, each sequence uses the "baseline-stimulus-baseline-stimulus-baseline -stimulus-baseline-stimulus-baseline-stimulus-baseline-stimulus-baseline-stimulus-baseline" model. The first baseline duration is 24s. The following baseline duration and duration of stimulus are 18s, each sequence is 240s, a total of three sequences. Scan 12min. From the Snodgrass picture database, 54 animal pictures and 54 tool pictures can be accurately identified by all subjects. Repeat 6 animal chunk and 6 tool naming chunks, six pictures of each block for 18 seconds. Choose the abstract map of all the American skunk as the baseline map of the animal name, and select the simple arrow picture as the baseline map of the tool. In order to avoid repetition effect after practice, the pictures used in the design of MRI are not repeated in speech behavior assessment. At baseline, subjects were asked to identify the direction of the arrow image and the tail direction of the skunk by silently speaking "upright" or "inverted". The subjects received task familiarization training before testing to ensure that there was no meaningless picture naming in baseline tasks, but location judgment. The design of language task is based on the design of Damasio. In the task state of magnetic resonance scanning, the patient is required to read and name the silent images of the visual images. The visual information is written by the DMDX software, the picture is projected through the brain functional audio-visual stimulation system (SA-9900) to the screen, and the subjects are placed on the head line. The reflector on the circle is observed.

Resting-state fMRI：During the rest-state fMRI scan, no task instruction was given to the participates, and the participates were completely relaxing, closing their eyes, breathing calmly, keeping their head still, but could not fall asleep, tried to avoid any systematic thinking activities, scanning 8min.

Functional magnetic resonance data acquisition：Cranial scanning was performed using the HDX3.0Tesla superconducting magnetic resonance scanner of the US GE company. The 8 channel phased array head coil is the receiving coil, and the scanning sequence and parameters are as follows：

1. T1 structure imaging using FSPGR BRAVO sequence. The parameters included: time of repetition, 8.86 ms; time of echo, 3.52 ms; field of view, 24×24 cm2; in-plane resolution,256×256; slice thickness, 1 mm;interslice gap, 1 mm; and number of slices, 176.
2. Echo-Planar Imaging (EPI) was used to acquire task-state fMRI data.The parameters included: time of repetition, 3000ms; time of echo, 40 ms; field of view, 24×24 cm2; in-plane resolution,64×64; slice thickness, 4 mm; interslice gap, 1 mm; and number of slices, 34. Scan a sequence of 240s, a total of 12 min.
3. Echo-Planar Imaging (EPI) was used to acquire rest-state fMRI data.The parameters included: time of repetition, 3000ms; time of echo, 40 ms; field of view, 24×24 cm2; in-plane resolution,64×64; slice thickness, 4 mm; interslice gap, 1 mm; and number of slices, 34. A total of 8 min.

ELIGIBILITY:
Inclusion Criteria:

* The first stroke of the left single subcortical areas, within 72hours.
* Primary school or higher level,aged between 18-75, native language Chinese
* According to the commonly used eye chart examination, the corrected visual acuity is more than 1.0.
* According to the Edinburgh Handedness Questionnaire (EHQ) as the right handed.
* The language function was normal before the onset. After the onset, the language function was mildly to moderately impaired with Western Aphasia Battery (WAB) ( Aphasia Quotient (AQ) between in 60 to 88).
* The patient cooperate with the examination, they and their guardian signed the informed consent

Exclusion Criteria:

* History of organic diseases of the nervous system and history of craniocerebral trauma.
* History of epilepsy and psychosis.
* History of material dependence.
* Decompensation of important organ function.
* Hamilton Depression Scale(HAMD )>8 points.
* Hamilton Anxiety Scale(HAMA )>7 points.
* The Mini-Mental State Examination (MMSE)score <20 points.
* Pregnant women and breast-feeding women.
* Contraindication of MRI scanning.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first onset, the onset time was less than 3 days, the lesion was the left and right single subcortical infarct lesion confirmed by head Magnetic Resonance Imaging(MRI).All of them are come from Neurology/Cerebrovascular Department General Hospital of Guangzhou Military Command of PLA between 2016-2017.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2016-10-09 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
A change of outcome measure: the Chinese version of Western Aphasia Battery(WAB) | This is an outcome measure to assess the improvement of language function from onset to 3 months after treatment. Thus, participates will undergo this assessment within 3 days (V1), 28±3 days (V2), and 90±3 days(V3) after randomization.
  The main outcome measure for this scale is Aphasia Quotient(AQ) which mainly tests the ability of spontaneous speech, oral comprehension, repetition, and naming, and reflects the severity of aphasia, and can be used as a reliable indicator to evaluate the improvement and deterioration of aphasia. Score fluctuation is 0-100 points, the normal value is 98.4-100 points, AQ<93.8 can be judged as language dysfunction.

SECONDARY OUTCOMES:
A change of outcome measure: Spontaneous Language Frequency Test(SLFT) | This is an outcome measure to assess the improvement of language function from onset to 3 months after treatment. Thus, participates will undergo this assessment within 3 days (V1), 28±3 days (V2), and 90±3 days(V3) after randomization.
  This test mainly assesses spontaneous speech fluency of participants. It requires participants name as many food names as possible within one minute, and each correct one to give one point. The higher the score, the better the language function.
A change of outcome measure: Picture Naming Test(PNT) | This is an outcome measure to assess the improvement of language function from onset to 3 months after treatment. Thus, participates will undergo this assessment on the within 3 days (V1), 28±3 days (V2), and 90±3 days(V3) after randomization.
  This test mainly assesses the ability of picture name of participants. we used a program for displaying named pictures on a computer screen (60 photos in total, of which 20 were Chinese celebrity faces). Each image was displayed in 3 seconds, and 1 point was correctly named for an image. The faces of celebrities were selected from the picture database of Chinese celebrities in the State Key Laboratory of Cognitive Neuroscience and Learning at Beijing Normal University. Score fluctuation is 0-60 points, the higher the score, the better the ability of picture name.
Follow-up measurement:Functional Magnetic Resonance Imaging(fMRI) | This is an outcome measure to assess the improvement of language function from onset to 3 months after treatment. Thus, participates will undergo this assessment within 3 days (V1), 28±3 days (V2), and 90±3 days(V3) after randomization.
  The examine included task-state fMRI and resting-state fMRI Time Frame: We will explore the mechanisms of dynamic changes in language functions. Thus, participates will undergo this examine on the first days (V1), 28±3 days (V2), and 90±3 days (V3) after randomization..

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yan, PhD, Study Chair — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Cerebrovascular Department of General Hospital of Guangzhou Military Command of PLA, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pedersen PM, Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Aphasia in acute stroke: incidence, determinants, and recovery. Ann Neurol. 1995 Oct;38(4):659-66. doi: 10.1002/ana.410380416. PMID 7574464
- [Background] Berthier ML. Poststroke aphasia : epidemiology, pathophysiology and treatment. Drugs Aging. 2005;22(2):163-82. doi: 10.2165/00002512-200522020-00006. PMID 15733022
- [Background] Engelter ST, Gostynski M, Papa S, Frei M, Born C, Ajdacic-Gross V, Gutzwiller F, Lyrer PA. Epidemiology of aphasia attributable to first ischemic stroke: incidence, severity, fluency, etiology, and thrombolysis. Stroke. 2006 Jun;37(6):1379-84. doi: 10.1161/01.STR.0000221815.64093.8c. Epub 2006 May 11. PMID 16690899
- [Background] Pizzamiglio L, Galati G, Committeri G. The contribution of functional neuroimaging to recovery after brain damage: a review. Cortex. 2001 Feb;37(1):11-31. doi: 10.1016/s0010-9452(08)70555-0. PMID 11292157
- [Background] Fridriksson J, Holland AL, Coull BM, Plante E, Trouard TP, Beeson P. Aphasia severity: Association with cerebral perfusion and diffusion. Aphasiology. 2002 Sep 1;16(9):859-871. doi: 10.1080/02687030244000347. PMID 16823466
- [Background] Hillis AE, Kleinman JT, Newhart M, Heidler-Gary J, Gottesman R, Barker PB, Aldrich E, Llinas R, Wityk R, Chaudhry P. Restoring cerebral blood flow reveals neural regions critical for naming. J Neurosci. 2006 Aug 2;26(31):8069-73. doi: 10.1523/JNEUROSCI.2088-06.2006. PMID 16885220
- [Background] Seitz RJ, Azari NP, Knorr U, Binkofski F, Herzog H, Freund HJ. The role of diaschisis in stroke recovery. Stroke. 1999 Sep;30(9):1844-50. doi: 10.1161/01.str.30.9.1844. PMID 10471434
- [Background] Kwakkel G, Kollen B, Lindeman E. Understanding the pattern of functional recovery after stroke: facts and theories. Restor Neurol Neurosci. 2004;22(3-5):281-99. PMID 15502272
- [Background] Warburton E, Price CJ, Swinburn K, Wise RJ. Mechanisms of recovery from aphasia: evidence from positron emission tomography studies. J Neurol Neurosurg Psychiatry. 1999 Feb;66(2):155-61. doi: 10.1136/jnnp.66.2.155. PMID 10071093
- [Background] Szaflarski JP, Allendorfer JB, Banks C, Vannest J, Holland SK. Recovered vs. not-recovered from post-stroke aphasia: the contributions from the dominant and non-dominant hemispheres. Restor Neurol Neurosci. 2013;31(4):347-60. doi: 10.3233/RNN-120267. PMID 23482065
- [Background] Heiss WD, Kessler J, Thiel A, Ghaemi M, Karbe H. Differential capacity of left and right hemispheric areas for compensation of poststroke aphasia. Ann Neurol. 1999 Apr;45(4):430-8. doi: 10.1002/1531-8249(199904)45:43.0.co;2-p. PMID 10211466
- [Background] Rosen HJ, Petersen SE, Linenweber MR, Snyder AZ, White DA, Chapman L, Dromerick AW, Fiez JA, Corbetta MD. Neural correlates of recovery from aphasia after damage to left inferior frontal cortex. Neurology. 2000 Dec 26;55(12):1883-94. doi: 10.1212/wnl.55.12.1883. PMID 11134389
- [Background] Meinzer M, Flaisch T, Breitenstein C, Wienbruch C, Elbert T, Rockstroh B. Functional re-recruitment of dysfunctional brain areas predicts language recovery in chronic aphasia. Neuroimage. 2008 Feb 15;39(4):2038-46. doi: 10.1016/j.neuroimage.2007.10.008. Epub 2007 Oct 18. PMID 18096407
- [Background] Calvert GA, Brammer MJ, Morris RG, Williams SC, King N, Matthews PM. Using fMRI to study recovery from acquired dysphasia. Brain Lang. 2000 Feb 15;71(3):391-9. doi: 10.1006/brln.1999.2272. PMID 10716869
- [Background] Lazar RM, Marshall RS, Pile-Spellman J, Duong HC, Mohr JP, Young WL, Solomon RL, Perera GM, DeLaPaz RL. Interhemispheric transfer of language in patients with left frontal cerebral arteriovenous malformation. Neuropsychologia. 2000;38(10):1325-32. doi: 10.1016/s0028-3932(00)00054-3. PMID 10869575
- [Background] Thulborn KR, Carpenter PA, Just MA. Plasticity of language-related brain function during recovery from stroke. Stroke. 1999 Apr;30(4):749-54. doi: 10.1161/01.str.30.4.749. PMID 10187873
- [Background] Buckner RL, Corbetta M, Schatz J, Raichle ME, Petersen SE. Preserved speech abilities and compensation following prefrontal damage. Proc Natl Acad Sci U S A. 1996 Feb 6;93(3):1249-53. doi: 10.1073/pnas.93.3.1249. PMID 8577749
- [Background] Gold BT, Kertesz A. Right hemisphere semantic processing of visual words in an aphasic patient: an fMRI study. Brain Lang. 2000 Jul;73(3):456-65. doi: 10.1006/brln.2000.2317. PMID 10860566
- [Background] Ohyama M, Senda M, Kitamura S, Ishii K, Mishina M, Terashi A. Role of the nondominant hemisphere and undamaged area during word repetition in poststroke aphasics. A PET activation study. Stroke. 1996 May;27(5):897-903. doi: 10.1161/01.str.27.5.897. PMID 8623110
- [Background] Weiller C, Isensee C, Rijntjes M, Huber W, Muller S, Bier D, Dutschka K, Woods RP, Noth J, Diener HC. Recovery from Wernicke's aphasia: a positron emission tomographic study. Ann Neurol. 1995 Jun;37(6):723-32. doi: 10.1002/ana.410370605. PMID 7778845
- [Background] Butefisch CM, Kleiser R, Seitz RJ. Post-lesional cerebral reorganisation: evidence from functional neuroimaging and transcranial magnetic stimulation. J Physiol Paris. 2006 Jun;99(4-6):437-54. doi: 10.1016/j.jphysparis.2006.03.001. Epub 2006 May 24. PMID 16723211
- [Background] Lang N, Nitsche MA, Paulus W, Rothwell JC, Lemon RN. Effects of transcranial direct current stimulation over the human motor cortex on corticospinal and transcallosal excitability. Exp Brain Res. 2004 Jun;156(4):439-43. doi: 10.1007/s00221-003-1800-2. Epub 2004 Jan 24. PMID 14745467
- [Background] Shimizu T, Hosaki A, Hino T, Sato M, Komori T, Hirai S, Rossini PM. Motor cortical disinhibition in the unaffected hemisphere after unilateral cortical stroke. Brain. 2002 Aug;125(Pt 8):1896-907. doi: 10.1093/brain/awf183. PMID 12135979
- [Background] Saur D, Lange R, Baumgaertner A, Schraknepper V, Willmes K, Rijntjes M, Weiller C. Dynamics of language reorganization after stroke. Brain. 2006 Jun;129(Pt 6):1371-84. doi: 10.1093/brain/awl090. Epub 2006 Apr 25. PMID 16638796
- [Background] Naeser MA, Martin PI, Nicholas M, Baker EH, Seekins H, Helm-Estabrooks N, Cayer-Meade C, Kobayashi M, Theoret H, Fregni F, Tormos JM, Kurland J, Doron KW, Pascual-Leone A. Improved naming after TMS treatments in a chronic, global aphasia patient--case report. Neurocase. 2005 Jun;11(3):182-93. doi: 10.1080/13554790590944663. PMID 16006338
- [Background] Barwood CH, Murdoch BE, Whelan BM, Lloyd D, Riek S, O' Sullivan JD, Coulthard A, Wong A. Improved language performance subsequent to low-frequency rTMS in patients with chronic non-fluent aphasia post-stroke. Eur J Neurol. 2011 Jul;18(7):935-43. doi: 10.1111/j.1468-1331.2010.03284.x. Epub 2010 Dec 7. PMID 21138505
- [Background] Heiss WD, Karbe H, Weber-Luxenburger G, Herholz K, Kessler J, Pietrzyk U, Pawlik G. Speech-induced cerebral metabolic activation reflects recovery from aphasia. J Neurol Sci. 1997 Feb 12;145(2):213-7. doi: 10.1016/s0022-510x(96)00252-3. PMID 9094051
- [Background] Belliveau JW, Cohen MS, Weisskoff RM, Buchbinder BR, Rosen BR. Functional studies of the human brain using high-speed magnetic resonance imaging. J Neuroimaging. 1991 Feb;1(1):36-41. doi: 10.1111/jon19911136. PMID 10183948
- [Background] Cramer SC, Nelles G, Benson RR, Kaplan JD, Parker RA, Kwong KK, Kennedy DN, Finklestein SP, Rosen BR. A functional MRI study of subjects recovered from hemiparetic stroke. Stroke. 1997 Dec;28(12):2518-27. doi: 10.1161/01.str.28.12.2518. PMID 9412643
- [Background] Tremblay P, Dick AS. Broca and Wernicke are dead, or moving past the classic model of language neurobiology. Brain Lang. 2016 Nov;162:60-71. doi: 10.1016/j.bandl.2016.08.004. Epub 2016 Aug 30. PMID 27584714
- [Background] Geschwind N. The organization of language and the brain. Science. 1970 Nov 27;170(3961):940-4. doi: 10.1126/science.170.3961.940. No abstract available. PMID 5475022
- [Background] Dick AS, Bernal B, Tremblay P. The language connectome: new pathways, new concepts. Neuroscientist. 2014 Oct;20(5):453-67. doi: 10.1177/1073858413513502. Epub 2013 Dec 15. PMID 24342910
- [Background] Rolston JD, Chang EF. Critical Language Areas Show Increased Functional Connectivity in Human Cortex. Cereb Cortex. 2018 Dec 1;28(12):4161-4168. doi: 10.1093/cercor/bhx271. PMID 29045564
- [Background] Buckner RL, Andrews-Hanna JR, Schacter DL. The brain's default network: anatomy, function, and relevance to disease. Ann N Y Acad Sci. 2008 Mar;1124:1-38. doi: 10.1196/annals.1440.011. PMID 18400922
- [Background] Foster BL, Dastjerdi M, Parvizi J. Neural populations in human posteromedial cortex display opposing responses during memory and numerical processing. Proc Natl Acad Sci U S A. 2012 Sep 18;109(38):15514-9. doi: 10.1073/pnas.1206580109. Epub 2012 Sep 4. PMID 22949666
- [Background] Andrews-Hanna JR. The brain's default network and its adaptive role in internal mentation. Neuroscientist. 2012 Jun;18(3):251-70. doi: 10.1177/1073858411403316. Epub 2011 Jun 15. PMID 21677128
- [Background] Chen Q, Beaty RE, Wei D, Yang J, Sun J, Liu W, Yang W, Zhang Q, Qiu J. Longitudinal Alterations of Frontoparietal and Frontotemporal Networks Predict Future Creative Cognitive Ability. Cereb Cortex. 2018 Jan 1;28(1):103-115. doi: 10.1093/cercor/bhw353. PMID 29253252
- [Background] Mancini S, Quinones I, Molinaro N, Hernandez-Cabrera JA, Carreiras M. Disentangling meaning in the brain: Left temporal involvement in agreement processing. Cortex. 2017 Jan;86:140-155. doi: 10.1016/j.cortex.2016.11.008. Epub 2016 Nov 18. PMID 27984788
- [Background] Crosson B. Thalamic mechanisms in language: a reconsideration based on recent findings and concepts. Brain Lang. 2013 Jul;126(1):73-88. doi: 10.1016/j.bandl.2012.06.011. Epub 2012 Jul 23. PMID 22831779
- [Background] Civier O, Bullock D, Max L, Guenther FH. Computational modeling of stuttering caused by impairments in a basal ganglia thalamo-cortical circuit involved in syllable selection and initiation. Brain Lang. 2013 Sep;126(3):263-78. doi: 10.1016/j.bandl.2013.05.016. Epub 2013 Jul 19. PMID 23872286
- [Background] Chai XJ, Berken JA, Barbeau EB, Soles J, Callahan M, Chen JK, Klein D. Intrinsic Functional Connectivity in the Adult Brain and Success in Second-Language Learning. J Neurosci. 2016 Jan 20;36(3):755-61. doi: 10.1523/JNEUROSCI.2234-15.2016. PMID 26791206
- [Background] Poeppel D, Emmorey K, Hickok G, Pylkkanen L. Towards a new neurobiology of language. J Neurosci. 2012 Oct 10;32(41):14125-31. doi: 10.1523/JNEUROSCI.3244-12.2012. PMID 23055482
- [Background] Catani M, Mesulam MM, Jakobsen E, Malik F, Martersteck A, Wieneke C, Thompson CK, Thiebaut de Schotten M, Dell'Acqua F, Weintraub S, Rogalski E. A novel frontal pathway underlies verbal fluency in primary progressive aphasia. Brain. 2013 Aug;136(Pt 8):2619-28. doi: 10.1093/brain/awt163. Epub 2013 Jul 2. PMID 23820597
- [Background] Broce I, Bernal B, Altman N, Tremblay P, Dick AS. Fiber tracking of the frontal aslant tract and subcomponents of the arcuate fasciculus in 5-8-year-olds: Relation to speech and language function. Brain Lang. 2015 Oct;149:66-76. doi: 10.1016/j.bandl.2015.06.006. Epub 2015 Jul 14. PMID 26186231
- [Background] Herrera-Guzman I, Herrera-Abarca JE, Gudayol-Ferre E, Herrera-Guzman D, Gomez-Carbajal L, Pena-Olvira M, Villuendas-Gonzalez E, Joan GO. Effects of selective serotonin reuptake and dual serotonergic-noradrenergic reuptake treatments on attention and executive functions in patients with major depressive disorder. Psychiatry Res. 2010 May 30;177(3):323-9. doi: 10.1016/j.psychres.2010.03.006. Epub 2010 Apr 10. PMID 20385412
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Damasio H, Grabowski TJ, Tranel D, Hichwa RD, Damasio AR. A neural basis for lexical retrieval. Nature. 1996 Apr 11;380(6574):499-505. doi: 10.1038/380499a0. PMID 8606767
- [Background] Beaulieu C, Allen PS. Determinants of anisotropic water diffusion in nerves. Magn Reson Med. 1994 Apr;31(4):394-400. doi: 10.1002/mrm.1910310408. PMID 8208115
- [Background] Alnaes D, Kaufmann T, Doan NT, Cordova-Palomera A, Wang Y, Bettella F, Moberget T, Andreassen OA, Westlye LT. Association of Heritable Cognitive Ability and Psychopathology With White Matter Properties in Children and Adolescents. JAMA Psychiatry. 2018 Mar 1;75(3):287-295. doi: 10.1001/jamapsychiatry.2017.4277. PMID 29365026
- [Background] Ganzola R, McIntosh AM, Nickson T, Sprooten E, Bastin ME, Giles S, Macdonald A, Sussmann J, Duchesne S, Whalley HC. Diffusion tensor imaging correlates of early markers of depression in youth at high-familial risk for bipolar disorder. J Child Psychol Psychiatry. 2018 Aug;59(8):917-927. doi: 10.1111/jcpp.12879. Epub 2018 Feb 28. PMID 29488219
- [Background] Dillon DG, Gonenc A, Belleau E, Pizzagalli DA. Depression is associated with dimensional and categorical effects on white matter pathways. Depress Anxiety. 2018 May;35(5):440-447. doi: 10.1002/da.22734. Epub 2018 Feb 27. PMID 29486093
- [Background] Basser PJ, Mattiello J, LeBihan D. MR diffusion tensor spectroscopy and imaging. Biophys J. 1994 Jan;66(1):259-67. doi: 10.1016/S0006-3495(94)80775-1. PMID 8130344
- [Background] Basser PJ, Jones DK. Diffusion-tensor MRI: theory, experimental design and data analysis - a technical review. NMR Biomed. 2002 Nov-Dec;15(7-8):456-67. doi: 10.1002/nbm.783. PMID 12489095
- [Background] Basser PJ, Pajevic S, Pierpaoli C, Duda J, Aldroubi A. In vivo fiber tractography using DT-MRI data. Magn Reson Med. 2000 Oct;44(4):625-32. doi: 10.1002/1522-2594(200010)44:43.0.co;2-o. PMID 11025519
- [Background] Lim JC, Phal PM, Desmond PM, Nichols AD, Kokkinos C, Danesh-Meyer HV, Kaye AH, Moffat BA. Probabilistic MRI tractography of the optic radiation using constrained spherical deconvolution: a feasibility study. PLoS One. 2015 Mar 5;10(3):e0118948. doi: 10.1371/journal.pone.0118948. eCollection 2015. PMID 25742640
- [Background] Theisen F, Leda R, Pozorski V, Oh JM, Adluru N, Wong R, Okonkwo O, Dean DC 3rd, Bendlin BB, Johnson SC, Alexander AL, Gallagher CL. Evaluation of striatonigral connectivity using probabilistic tractography in Parkinson's disease. Neuroimage Clin. 2017 Sep 9;16:557-563. doi: 10.1016/j.nicl.2017.09.009. eCollection 2017. PMID 28971007
- [Background] Galantucci S, Tartaglia MC, Wilson SM, Henry ML, Filippi M, Agosta F, Dronkers NF, Henry RG, Ogar JM, Miller BL, Gorno-Tempini ML. White matter damage in primary progressive aphasias: a diffusion tensor tractography study. Brain. 2011 Oct;134(Pt 10):3011-29. doi: 10.1093/brain/awr099. Epub 2011 Jun 11. PMID 21666264
- [Background] Kim H, Na DL. Normative data on the Korean version of the Western Aphasia Battery. J Clin Exp Neuropsychol. 2004 Nov;26(8):1011-20. doi: 10.1080/13803390490515397. PMID 15590457
- [Background] Xie Q, Liu Y, Li CY, Song XZ, Wang J, Han LX, Bai HM. The modulation of venlafaxine on cortical activation of language area in healthy subjects with fMRI study. Psychopharmacology (Berl). 2012 Oct;223(4):417-25. doi: 10.1007/s00213-012-2730-0. Epub 2012 May 4. PMID 22555622
- [Background] Oguz I, Farzinfar M, Matsui J, Budin F, Liu Z, Gerig G, Johnson HJ, Styner M. DTIPrep: quality control of diffusion-weighted images. Front Neuroinform. 2014 Jan 30;8:4. doi: 10.3389/fninf.2014.00004. eCollection 2014. PMID 24523693
- [Background] Andersson JLR, Sotiropoulos SN. An integrated approach to correction for off-resonance effects and subject movement in diffusion MR imaging. Neuroimage. 2016 Jan 15;125:1063-1078. doi: 10.1016/j.neuroimage.2015.10.019. Epub 2015 Oct 20. PMID 26481672